CLINICAL TRIAL: NCT02838095
Title: Effectiveness of a Daytime Nap on Alleviating Cognitive Impairment Due to Short Sleep in Adolescents
Brief Title: Effects of Napping in Sleep-Restricted Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke-NUS Graduate Medical School (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Principal Investigator, Michael WL Chee, MBBS, Professor, Neuroscience and Behavioural Disorders Program; Director, Centre for Cognitive Neuroscience, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NFS2
Record Dates: First submitted 2016-06-15; First posted 2016-07-20 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Sleep Deprivation; Sleep
Keywords: nap; sleep restriction; recovery sleep; cognitive performance; subjective sleepiness; mood; neurobehavioural functions
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No nap (No Intervention): After each night with a 5-hour sleep opportunity, participants did not have a daytime nap opportunity, but instead watched documentaries.
- Nap (Experimental): After each night with a 5-hour sleep opportunity, participants had the chance to take a daytime nap from 14:00 to 15:00.
  Interventions: Behavioral: Nap

INTERVENTIONS:
Behavioral: Nap — A 1-hour daytime nap opportunity
  Arms: Nap

SUMMARY:
To examine the neurobehavioural responses to two successive cycles of sleep restriction and recovery in adolescents, and to determine the benefits of napping on cognitive performance, alertness, and mood. 57 participants, aged 15 to 19 years old, were divided into nap and no-nap groups. Both groups underwent two cycles of sleep restriction and recovery over 15 days. The nap group received an afternoon sleep opportunity lasting 1 hour.

DETAILED DESCRIPTION:
57 participants (aged 15 to 19 years old) were grouped into nap and no nap groups. Both groups took part in a 15-day protocol that started with 2 9-hour adaptation and baseline nights, followed by two successive cycles of sleep restriction (5-h time-in-bed [TIB]; 01:00-06:00) and recovery (9-h TIB; 23:00-08:00) intended to simulate the weekday sleep loss and weekend attempt to 'catch up' that are familiar to high school students. The nap group received a 1-hour nap opportunity at 14:00 following each sleep-restricted night, while participants in the no nap group watched a documentary. Sleep was monitored with polysomnography on 9 selected nights. Cognitive performance, subjective sleepiness, and mood were assessed 3 times daily (10:00, 15:45, and 20:00).

All participants stayed in air-conditioned, twin-share bedrooms with en-suite bathrooms. Bedroom windows were fitted with blackout panels to ensure participants were not woken up prematurely by sunlight. Earplugs were also provided, and participants were allowed to adjust the temperature of their bedrooms to their personal comfort. 3 main meals were served each day, with snacks being provided for upon request. Caffeinated drinks, unscheduled sleep, and strenuous physical activities were prohibited.

Outside of scheduled sleep, meal, and cognitive testing times, participants spent the majority of their free time in a common room that was illuminated by natural and artificial lighting. They were allowed to read, play non-physically exerting games, watch videos, and interact with research staff and other participants. Participants were under constant supervision by the research staff.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* no sleep disorder
* body mass index not greater than 30

Exclusion Criteria:

* smoker
* habitual short sleeper (time in bed during term time of less than 6 hours and no sign of sleep extension of greater than 1 hour on weekends)
* consumption of more than 5 cups of caffeinated beverages a day
* travelling across more than 2 time zones in the month prior to the study protocol
* diagnosed with any psychiatric conditions

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 57 (Actual)
Dates: Start 2015-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in sustained attention assessed with the Psychomotor Vigilance Task from morning to afternoon and then evening from baseline days to the first and second cycles of sleep restriction and recovery | 3 times daily (10:00, 15:45, and 20:00) for 15 days
  Number of attention lapses (>500ms)
Change in working memory assessed with the 1-back task from morning to afternoon and then evening from baseline days to the first and second cycles of sleep restriction and recovery | 3 times daily (10:00, 15:45, and 20:00) for 15 days
  Number of correct responses in the 1-back task
Change in executive functions assessed with the 3-back task from morning to afternoon and then evening from baseline days to the first and second cycles of sleep restriction and recovery | 3 times daily (10:00, 15:45, and 20:00) for 15 days
  Number of correct responses in the 3-back task
Change in the level of subjective sleepiness assessed with the Karolinska Sleepiness Scale from morning to afternoon and then evening from baseline days to the first and second cycles of sleep restriction and recovery | 3 times daily (10:00, 15:45, and 20:00) for 15 days
  Score on the Karolinska Sleepiness Scale (1-9 points)
Change in positive mood assessed with the Positive and Negative Affect Scale (PANAS) from morning to afternoon and then evening from baseline days to the first and second cycles of sleep restriction and recovery | 3 times daily (10:00, 15:45, and 20:00) for 15 days
  Total score on the positive subscale of the PANAS
Change in negative mood assessed with the Positive and Negative Affect Scale (PANAS) from morning to afternoon and then evening from baseline days to the first and second cycles of sleep restriction and recovery | 3 times daily (10:00, 15:45, and 20:00) for 15 days
  Total score on the negative subscale of the PANAS
Change in speed of processing assessed with the Mental Arithmetic Task from morning to afternoon and then evening from baseline days to the first and second cycles of sleep restriction and recovery | 3 times daily (10:00, 15:45, and 20:00) for 15 days
  Number of correct responses in the task
Change in speed of processing assessed with the Symbol Digit Modalities Task from morning to afternoon and then evening from baseline days to the first and second cycles of sleep restriction and recovery | 3 times daily (10:00, 15:45, and 20:00) for 15 days
  Number of correct responses in the task

SECONDARY OUTCOMES:
Change in total sleep duration at night assessed with polysomnography from baseline nights to the first and second cycles of sleep restriction and recovery | Nocturnal sleep on nights 1 & 3 (baseline), 4, 6 & 8 (first sleep restriction period), 9 (first recovery period), 11 & 13 (second sleep restriction period), & 14 (second recovery period)
  Total duration of nocturnal sleep was determined to establish baseline sleep characteristics (first and third nights) and changes in the first sleep restriction period (fourth, sixth and eighth night), the first recovery period (ninth night), the second sleep restriction period (eleventh and thirteenth night), and the second recovery period (fourteenth night).
Change in N1 sleep duration at night assessed with polysomnography from baseline nights to the first and second cycles of sleep restriction and recovery | Nocturnal sleep on nights 1 & 3 (baseline), 4, 6 & 8 (first sleep restriction period), 9 (first recovery period), 11 & 13 (second sleep restriction period), & 14 (second recovery period)
  Duration of nocturnal N1 sleep was determined to establish baseline sleep characteristics (first and third nights) and changes in the first sleep restriction period (fourth, sixth and eighth night), the first recovery period (ninth night), the second sleep restriction period (eleventh and thirteenth night), and the second recovery period (fourteenth night).
Change in N2 sleep duration at night assessed with polysomnography from baseline nights to the first and second cycles of sleep restriction and recovery | Nocturnal sleep on nights 1 & 3 (baseline), 4, 6 & 8 (first sleep restriction period), 9 (first recovery period), 11 & 13 (second sleep restriction period), & 14 (second recovery period)
  Duration of nocturnal N2 sleep was determined to establish baseline sleep characteristics (first and third nights) and changes in the first sleep restriction period (fourth, sixth and eighth night), the first recovery period (ninth night), the second sleep restriction period (eleventh and thirteenth night), and the second recovery period (fourteenth night).
Change in N3 sleep duration at night assessed with polysomnography from baseline nights to the first and second cycles of sleep restriction and recovery | Nocturnal sleep on nights 1 & 3 (baseline), 4, 6 & 8 (first sleep restriction period), 9 (first recovery period), 11 & 13 (second sleep restriction period), & 14 (second recovery period)
  Duration of nocturnal N3 sleep was determined to establish baseline sleep characteristics (first and third nights) and changes in the first sleep restriction period (fourth, sixth and eighth night), the first recovery period (ninth night), the second sleep restriction period (eleventh and thirteenth night), and the second recovery period (fourteenth night).
Change in REM sleep duration at night assessed with polysomnography from baseline nights to the first and second cycles of sleep restriction and recovery | Nocturnal sleep on nights 1 & 3 (baseline), 4, 6 & 8 (first sleep restriction period), 9 (first recovery period), 11 & 13 (second sleep restriction period), & 14 (second recovery period)
  Duration of nocturnal REM sleep was determined to establish baseline sleep characteristics (first and third nights) and changes in the first sleep restriction period (fourth, sixth and eighth night), the first recovery period (ninth night), the second sleep restriction period (eleventh and thirteenth night), and the second recovery period (fourteenth night).
Change in total sleep duration during daytime naps assessed with polysomnography from the first to the second sleep restriction period | Afternoon naps on days 4, 6 & 8 (first sleep restriction period), 11 & 13 (second sleep restriction period)
  Total duration of sleep during the selected nap episodes was determined to track changes in this parameter from the first sleep restriction period (fourth, sixth and eighth day) to the second sleep restriction period (eleventh and thirteenth day).
Change in N1 sleep duration during daytime naps assessed with polysomnography from the first to the second sleep restriction period | Afternoon naps on days 4, 6 & 8 (first sleep restriction period), 11 & 13 (second sleep restriction period)
  Duration of N1 sleep during the selected nap episodes was determined to track changes in this parameter from the first sleep restriction period (fourth, sixth and eighth day) to the second sleep restriction period (eleventh and thirteenth day).
Change in N2 sleep duration during daytime naps assessed with polysomnography from the first to the second sleep restriction period | Afternoon naps on days 4, 6 & 8 (first sleep restriction period), 11 & 13 (second sleep restriction period)
  Duration of N2 sleep during the selected nap episodes was determined to track changes in this parameter from the first sleep restriction period (fourth, sixth and eighth day) to the second sleep restriction period (eleventh and thirteenth day).
Change in N3 sleep duration during daytime naps assessed with polysomnography from the first to the second sleep restriction period | Afternoon naps on days 4, 6 & 8 (first sleep restriction period), 11 & 13 (second sleep restriction period)
  Duration of N3 sleep during the selected nap episodes was determined to track changes in this parameter from the first sleep restriction period (fourth, sixth and eighth day) to the second sleep restriction period (eleventh and thirteenth day).
Change in REM sleep duration during daytime naps assessed with polysomnography from the first to the second sleep restriction period | Afternoon naps on days 4, 6 & 8 (first sleep restriction period), 11 & 13 (second sleep restriction period)
  Duration of REM sleep during the selected nap episodes was determined to track changes in this parameter from the first sleep restriction period (fourth, sixth and eighth day) to the second sleep restriction period (eleventh and thirteenth day).

CONTACTS AND LOCATIONS:
Overall Officials: Michael WL Chee, MBBS, Principal Investigator — Duke-NUS Graduate Medical School
Locations (1):
- Duke-NUS Medical School, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lo JC, Ang JWA, Koa TB, Ong JL, Lim J. Predicting vigilance vulnerability during 1 and 2 weeks of sleep restriction with baseline performance metrics. Sleep Adv. 2022 Oct 25;3(1):zpac040. doi: 10.1093/sleepadvances/zpac040. eCollection 2022. PMID 37193393
- [Derived] Lo JC, Koa TB, Ong JL, Gooley JJ, Chee MWL. Staying vigilant during recurrent sleep restriction: dose-response effects of time-in-bed and benefits of daytime napping. Sleep. 2022 Apr 11;45(4):zsac023. doi: 10.1093/sleep/zsac023. PMID 35089345